CLINICAL TRIAL: NCT01850147
Title: Study of Efficacy and Safety of Sequential Low-dose Sunitinib With Chemotherapy in Advanced Non-small Cell Lung Cancer After Failure of Conventional Regimen
Brief Title: Sequential Use of Low-dose Sunitinib With Chemotherapy in Advanced NSCLC After Failure of Conventional Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LI Junling, Professor and Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-2013-041
Record Dates: First submitted 2013-04-18; First posted 2013-05-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Cancer; Lung Cancer
Keywords: sunitinib; chemotherapy; non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Sunitinib; Drug Therapy

ARMS (1):
- Sunitinib (Experimental)
  Interventions: Drug: Sunitinib, chemotherapy

INTERVENTIONS:
Drug: Sunitinib, chemotherapy — sunitinib, 12.5mg/day, for 7 days before each cycle of chemotherapy; chemotherapy, single agent including docetaxel, albumin-bound paclitaxel, vinorelbine, gemcitabine, pemetrexed, or paclitaxel, as determined by the investigator

SUMMARY:
The purpose of this study is to determine whether sequential application of low-dose short-term sunitinib and chemotherapy is effective in the treatment of non-small cell lung cancer after failure of conventional therapy. Safety of this regimen will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of stage IIIB/IV NSCLC
* ECOG PS: 0,1
* Unidimensional or bi-dimensional measurable disease
* Receive prior treatment including first-line platinum-based chemotherapy, standard second-line chemotherapy and 1 EGF/EGFR inhibitor
* Evidence of disease progression
* Life expectancy >12 weeks
* Neutrophils > 1.5 109/l, Platelets > 100 109/l, Hemoglobin > 9g/dl, Total bilirubin < 1.5 UNL, AST (SGOT) and ALT (SGPT) < 2.5 UNL, Alkaline phosphatases < 5 UNL, Creatinine < 1 UNL

Exclusion Criteria:

* Pre-existing hemoptysis of a severity > grade 3 by NCI CTCAE criteria within 4 weeks prior to study entry
* Uncontrolled hypertension
* CHF, angina or arrhythmias
* LVEF < 1 UNL
* Existing a second malignancy within 5 years
* Infected with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | up to 2 years
  The primary objective of this study is to evaluate the median progression-free survival of this sequential regimen.

SECONDARY OUTCOMES:
overall survival | up to 2 years
  To evaluate the median over-all survival of this regimen
disease control rate | up to 6 months
  To evaluate the disease-control rate of this regimen.
Safety | up to 2 years
  To evaluate the safety of this regimen including the rate and grade of adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China